CLINICAL TRIAL: NCT01797822
Title: Effects of Conventional Dry Eye Treatments on the Ocular Surface Response to Low Humidity Environment in Patients With Keratoconjunctivitis Sicca.
Brief Title: Effects of Dry Eye Treatments on the Ocular Surface
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Steven Pflugfelder, Professor of Ophthalmology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-31756
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Keratoconjunctivitis Sicca; Dry Eye Syndrome
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — Dexamethasone; Adrenal Cortex Hormones; Lubricant Eye Drops

STUDY DESIGN:
Masking Description: Vehicle and therapy groups were not masked.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artificial tears first, then Dexamethasone (Experimental): Artificial tears four times a day both eyes for two weeks, then Dexamethasone 0.01% four times a day both eyes for two weeks
  Interventions: Drug: Dexamethasone; Drug: Artificial tear

INTERVENTIONS:
Drug: Dexamethasone
  Other Names: corticosteroid, vehicle
Drug: Artificial tear

SUMMARY:
The purpose of this study is to evaluate whether, in people with dry eye syndrome, over the counter artificial tears and the prescription eye drop, dexamethasone, change or effect the eyes response to a low humidity environment.

It is known that irritation from dry eye can be improved by over the counter artificial tears because they wet and lubricate the eyes. The prescription eye drop, dexamethasone, can also improve eye irritation by decreasing the inflammation that develops in dry eye. Thus, the investigators hypothesize that the use of these conventional dry eye treatments will improve the eyes' response to a low humidity environment.

DETAILED DESCRIPTION:
This study evaluated the effects of the corticosteroid dexamethasone on suppressing development of eye irritation, cornea epithelial disease and increased production of inflammatory mediators in subjects who were subjected to an experimental low humidity drafty environment.

ELIGIBILITY:
Inclusion Criteria:

* Signature on the written informed consent form
* Patient motivation and willingness to cooperate with the investigator by following the required medication regimen
* Patient willingness and ability to return for all visits during the study
* Rapid tear film break up time of seven seconds or less in at least one eye AND
* Both cornea fluorescein staining score 3 or greater and conjunctival lissamine green staining 3 or greater in at least one eye
* Ocular Surface Disease Index Symptom Severity score of twenty or greater
* Tear meniscus height less than or equal to 200um
* Intact corneal sensitivity
* Willingness to discontinue use of any current dry eye treatment (except artificial tears) for four weeks prior to enrollment, and during the course of the study

Exclusion Criteria:

* Compromised cognitive ability which may be expected to interfere with study compliance
* Uncontrolled or poorly controlled diabetes or heart or pulmonary disease that could, in the judgment of the investigator, jeopardize subject safety or interfere with the interpretation of the results of the study
* Known hypersensitivity to any components of the artificial tears or dexamethasone eye drops
* Anticipated contact lens wear during the study
* History of corneal transplant
* Active ocular infection, uveitis or non-Keratoconjunctivitis sicca related inflammation
* History of cataract surgery within 3 months prior to enrollment
* History of pterygium removal within 6 months prior to enrollment
* Reduced corneal sensitivity
* Initiation, discontinuation or change in dosage of hormone replacement therapy, fish oil, evening primrose, flaxseed, or black current seed oil supplements, antihistamines, cholinergic agents, beta-blocking agents, tricyclic or selective serotonin reuptake inhibitors, antidepressants, phenothiazines, or topical or systemic acne rosacea medications in two months prior to enrollment, or anticipated change in dosage during course of study
* Topical ophthalmic medications within prior 4 weeks, or anticipated use of same during the study (except artificial tears)
* Occlusion of the lacrimal puncta either surgically or with temporary collagen punctal plugs within three months prior to study, or anticipated use of same during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pflugfelder, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Alkek Eye Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data was published in a peer reviewed publication
Supporting Information: Study Protocol
Time Frame: data is available in a peer reviewed publication
Access Criteria: data is available in a peer reviewed publication

RESULTS

PARTICIPANT FLOW:
Groups:
- Artificial Tears First, Then Dexamethasone 0.01%: Artificial tears four times a day for two weeks in both eyes, then Dexamethasone 0.01% ophthalmic solution four times a day for two weeks in both eyes
Period: Overall Study
Arm/Group | Artificial Tears First, Then Dexamethasone 0.01%
Started | 20
Completed | 20 (The protocol is now closed.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Dexamethasone, Artificial Tears: Dexamethasone 0.01% ophthalmic solution four times a day for two weeks in both eyes Artificial tears four times a day for two weeks in both eyes
  dexamethasone, artificial tears
Arm/Group | Dexamethasone, Artificial Tears
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.25 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Corneal Fluorescein Staining
Description: Subjects will be treated with preservative-free artificial tears for 2 weeks then exposed to a low humidity environment for 90 minutes, then treated with preservative-free dexamethasone 0.1% for 2 weeks and exposed to a low humidity environment again. The change in corneal fluorescein staining before and after the low humidity exposure was measured after each treatment. Fluorescein staining was graded using the CCLR scale (0-100) in 5 zones on the cornea for a maximum score of 500 (range 0-500). A lower change in staining indicates less severe disease in response to the low humidity stress. Negative number indicates staining after exposure was lower than pre.
Time Frame: Two weeks after treatment and exposure to a low humidity environment
Population: difference (change) in fluorescein staining pre- and post-exposure to low humidity stress
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Artificial Tears: Artificial tears four times a day for two weeks in both eyes/Artificial tears
- Dexamethasone: Dexamethasone 4 times per day for 2 weeks in both eyes/Dexamethasone
Arm/Group | Artificial Tears | Dexamethasone
Number analyzed (Participants) | 20 | 20
units on a scale | 22.18 (22.03) | -3.35 (18.83)
Statistical Analysis 1: Comparison: Artificial Tears vs Dexamethasone; Test type: Other — Statistical comparison between groups was made with t-test. A sample size of 20 subjects was calculates to have 90% power of detecting a statistical difference (P<0.05) in change in corneal staining pre and post low humidity challenge; p < 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Dexamethasone: Dexamethasone 0.01% ophthalmic solution four times a day for two weeks in both eyes
- Artificial Tear: Artificial tears four times a day for two weeks in both eyes
Arm/Group | Dexamethasone | Artificial Tear
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes